CLINICAL TRIAL: NCT04348266
Title: Efficacy of Radiofrequency Ablation in Treatment of Gastric Intestinal Metaplasia: a Randomized, Self-control Study
Brief Title: RFA for GIM Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Principle investigator, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP020
Record Dates: First submitted 2020-04-12; First posted 2020-04-16 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Gastric Intestinal Metaplasia; Treatment; Radio-frequency Ablation
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Study in only GIM patients but will divide the stomach into 2 sites (left and right) to random for RFA treatment.
Who Masked: Outcomes Assessor
Masking Description: The endoscopist who do the final endoscopy for assessing the efficacy of RFA will be blinded to the previous assigned location of RFA treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA (Experimental): The assigned location will be treated with RFA at all lesion.
  Interventions: Device: Radiofrequency ablation (RFA)
- Control (No Intervention): No treatment will not be performed at this location. However, if endoscopist detects any suspicious lesion during the scheduled endoscopy, the biopsy will be done and standard treatment will be performed accordingly.

INTERVENTIONS:
Device: Radiofrequency ablation (RFA) — Radiofrequency ablation is a device that can generate the heat from radiofrequency for tissue ablation. RFA is a standard treatment for Barrett' esophagus and high grade dysplasia in esophagus.
  Arms: RFA

SUMMARY:
Use radiofrequency ablation (RFA) for Gastric intestinal metaplasia (GIM) treatment.

DETAILED DESCRIPTION:
Gastric intestinal metaplasia (GIM) is a pre-malignant lesion. Currently, there is no standard treatment for this condition, thus the patients with GIM need surveillance endoscopy every 1-3 years, regarding to the severity and extension of lesion. However, the protocol for GIM surveillance is uncertain and need high cost.

Radiofrequency ablation (RFA) is used for Barrett's esophagus (BE; pre-malignant lesion of esophageal adenoCA) treatment as a standard treatment. The investigators hypothesized that RFA may effective in GIM treatment.

The investigators will random GIM participants to have the RFA treatment only one site of the stomach (left or right). At the first session, the investigators will biopsy at suspected GIM lesions to confirm the diagnosis and severity of GIM. Two months later, The investigators will apply RFA to all GIM lesions at the assigned location and then every 2 months for 3 sessions or until no GIM lesion seen by endoscopy. The final endoscopy will be done at 1 year follow-up and biopsy will be performed to assess the efficacy of RFA compare to no treatment.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Previous diagnose of extensive or incomplete GIM

Exclusion Criteria:

* No GIM at first endoscopy
* Previous gastric surgery
* Coagulopathy
* Pregnancy or lactation
* Unable to perform appropriate peri-procedural cessation of antiplatelet/antithrombotic therapy
* Unable to sign the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of GIM lesions regression | 1 year
  Regression of GIM lesions after RFA treatment compared to no treatment

SECONDARY OUTCOMES:
Number of GIM regression by location | 1 year
  Regression from extensive to non-extensive GIM after RFA treatment compared to no treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Rapat Pittayanon, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Do not share IPD to other researchers